CLINICAL TRIAL: NCT01998347
Title: Paclitaxel Liposome and Cisplatin as First-line Chemotherapy in Patients With Metastatic Esophageal Cancer: an Open-label, Randomised Phase 3 Trial.
Brief Title: Paclitaxel Liposome and Cisplatin as First-line Chemotherapy in Patients With Metastatic Esophageal Cancer
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: slow enrollment
Sponsor: Shantou University Medical College (Other)
Responsible Party: Principal Investigator, Lin Yingcheng, deputy secretary, Shantou University Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSMECS 01; LYC01 (Other: ShantouUMC)
Record Dates: First submitted 2013-11-17; First posted 2013-11-28 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paclitaxel liposome and Cisplatin (Experimental): Drug: paclitaxel liposome 175mg/m2, IV (in the vein) on day 1 of each 21 day cycle. Number of Cycles:up to 6 cycles.
  Drug: cisplatin 37.5 mg/m2, IV (in the vein) on day 1~2 of each 21 day cycle. Number of Cycles: up to 6 cycles.
  Interventions: Drug: Paclitaxel liposome; Drug: Cisplatin
- Cisplatin plus 5-fluorouracil (Active Comparator): Cisplatin:
  37.5 mg/m2, IV (in the vein) on day 1-2 of each 21 day cycle. Number of Cycles: up to 6 cycles.
  5-fluorouracil: 200mg/m2, CIV (continuous intravenous infusion) on day 1~5 of each 21 day cycle. Number of Cycles: up to 6 cycles.
  Interventions: Drug: Cisplatin; Drug: 5-fluorouracil

INTERVENTIONS:
Drug: Paclitaxel liposome
  Arms: Paclitaxel liposome and Cisplatin
Drug: Cisplatin
Drug: 5-fluorouracil
  Arms: Cisplatin plus 5-fluorouracil

SUMMARY:
There are no standard chemotherapy regimens for metastatic esophageal cancer. Cisplatin plus 5-fluorouracil is widely used as first-line treatment with a response rate ranged from 30% to 40%. Combination of paclitaxel and cisplatin has been investigated in small size clinical trial, producing promising outcome.Liposome capsuled paclitaxel has been proved to be as effective as paclitaxel.The usefulness of the the regimen of paclitaxel liposome with cisplatin is evaluated by median survival time, progression free survival,and response rate.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic esophageal tumors with no previous treatment for advanced disease or recurrent disease after previous treatment for at least one year.
* At least one measurable lesion according to the RECIST1.1 (Response Evaluation Criteria in Solid Tumors RECIST Version 1.1) criteria. Minimum indicator lesion size: > 10 mm measured by spiral CT or >20mm measured by conventional techniques.
* Patients aged between 18 and 70 years, inclusive, at the time of acquisition of informed consent
* Patients with performance status(ECOG) 0 to 1.
* Abnormal hematologic values (WBC ≥ 3.0 x 109/L, Hemoglobin ≥ 10.0g/dl, platelet count ≥ 100 x 109/L)
* Creatinine clearance ≥ 60 ml/min, Serum creatinine ≤ 1.5mg/dl
* Serum bilirubin ≤ 1.5mg/dl. ALT(Alanine transaminase ), AST(Aspartate Transaminase) ≤ 2.5 x upper normal limit (or ≤ 2.5 x upper normal limit in the case of liver metastases)
* Life expectancy ≥ 3 months
* Patients who have given written informed consent to participate in this study

Exclusion Criteria:

* Patients with active multiple cancers; or even if the multiple cancers are metachronous, have a disease-free period of less than 5 years (but excluding cancer in situ and skin cancer)
* Serious, uncontrolled, concurrent infection(s) or illness(es)
* Patients with no serious concurrent complications (such as heart disease, Intestinal pneumonia)
* Patients with brain metastasis
* Patients receiving continuous administration of steroids
* Patients who have experienced serious drug allergy in the past
* Patients with retention of body fluid(pleural effusion, ascites, pericardial effusion) necessitating treatment
* Patients who are pregnant and lactating or hope to become pregnant during the study period
* Patients with prior Taxane treatment (Paclitaxel)
* Others, patients judged by the investigator or coinvestigator to be inappropriate as subject

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-11; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
median overall survival | one year

SECONDARY OUTCOMES:
median progression free survival | 6 months

OTHER OUTCOMES:
time to progression | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of medical oncology,Cancer hospital of Shantou University Medical colledge, Shantou, Guangdong, China